CLINICAL TRIAL: NCT04257071
Title: Pilot Feasibility Study of Out-of-Pocket Cost Communication and Supportive Financial Services for Reducing Financial Toxicity Among Multiple Sclerosis Patients
Brief Title: Out of Pocket Cost Communication in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Gelareh Sadigh, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00113357
Record Dates: First submitted 2020-02-04; First posted 2020-02-05 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis
Keywords: Financial toxicity; Financial burden; Financial distress; Medical expense; Out of Pocket cost; Cost communication; Cost optimization; Price transparency; Financial navigation
MeSH Terms: conditions — Multiple Sclerosis; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Participants randomized to the usual care study arm will receive the usual care for their MS.
  Interventions: Behavioral: Usual Care
- OOP Cost Communication and Optimization (Experimental): Participants in this study arm in addition to usual care, will receive a personalized discussion of their OOP cost estimates for treatment obtained through an online price transparency tool, personalized analysis of expenses by financial counselor, and enrollment in any cost optimization opportunities for which they are eligible using a comprehensive financial navigation program.
  Interventions: Behavioral: Usual Care; Behavioral: OOP Cost Communication and Optimization

INTERVENTIONS:
Behavioral: Usual Care — The usual care for MS involves standard patient neurology visits and encounters with pharmacists, financial counselors and social workers if patients need any financial assistance with medication or other expenses.
Behavioral: OOP Cost Communication and Optimization — OOP Cost Communication and Optimization includes personalized discussion of OOP cost estimates for treatment plan obtained through an online price transparency tool, personalized analysis of patients' expenses by financial counselor, and patient enrollment in any cost optimization opportunities for which patient is eligible using a comprehensive financial navigation program.
  Arms: OOP Cost Communication and Optimization

SUMMARY:
This is a prospective randomized controlled trial of a cohort of adult multiple sclerosis (MS) patients visiting an outpatient neurology clinic. Sixty participants will be randomly assigned to the intervention arm or a control arm and will be followed for three months.

DETAILED DESCRIPTION:
Patients with multiple sclerosis (MS) spend a substantial amount on healthcare services (total lifetime cost of $4.1 million), and rank second behind congestive heart failure in direct all-cause medical costs for chronic conditions. Among medically bankrupt families, MS is reported to be associated with the highest out-of-pocket expenditure (mean $34,167) followed by diabetes, injuries, stroke, mental illness, and heart disease. With increased costs of MS disease-modifying therapies (DMTs) over the last 20 years, relatively higher out-of-pocket (OOP) costs for advanced imaging tests compared to other common essential health benefits, and increased cost sharing, the financial burden on MS patients continues to escalate. More than half of MS patients lose their ability to generate incomes within a decade after diagnosis due to disability. Accordingly, these patients are at high risk for health-related financial toxicity (a term used interchangeably with financial distress or financial burden, first introduced in the oncology literature to report potential economic impact of modern oncology medications). Financial toxicity is defined as a combination of subjective financial concerns (e.g., anxiety), objective financial consequences of health issues and treatments (e.g., decreased income, medical debt, bankruptcy), and patients' coping behaviors. Financial toxicity, as measured by the Comprehensive Score for Financial Toxicity Patient-Reported Outcome (COST), can harm patients' health-related quality of life (HRQOL). Further, the financial burden from high cost-sharing medical services can be a risk factor for treatment non-adherence. To date, there are no published studies measuring financial toxicity in MS patients, and work in other disease states cannot necessarily be generalized to MS patients. First, the economic burden of MS is different from cancer due to early age of disease onset and its progressive disabling course. Additionally, since MS affects people in the most productive stages of their lives, the disease additionally carries important social burdens.

Providing patients with resources to proactively manage the costs of their care may help to reduce financial toxicity. However, financial navigation, must be provided in a manner that is acceptable, accessible, less cumbersome, thereby not affecting the flow of clinical care. In order to better understand how to equip patients with tools that have the potential to reduce financial toxicity, there is an urgent need to study interventions at the patient, clinic, payer, and policy level.

This is a two-arm, randomized trial with 60 adult MS patients who are receiving disease modifying therapy to test the feasibility of OOP cost communication and optimization through centralized financial navigation and explore its efficacy to reduce financial toxicity and care non-adherence compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* known diagnosis of MS as documented in the electronic medical record by a neurologist based on clinical and imaging findings
* a prescription for DMTs as medication
* not enrolled in a clinical trial that covers the cost of DMT
* have capacity to consent

Exclusion Criteria:

* plan to receive treatment elsewhere
* concurrent diagnosis of primary cancers (except for non-melanoma skin cancer)
* unable to read and speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Questionnaire | Month 3
  Patient satisfaction with their experience with the OOP cost discussion and financial counselors is assessed with a 14-item Patient Satisfaction Questionnaire. Participants report how much they agree with each statement on a scale of 1 (strongly disagree) to 5 (strongly agree). Total scores range from 14 to 70 where higher scores indicate greater satisfaction with the financial counselor experiences.

SECONDARY OUTCOMES:
Percentage of Patients Participating in Cost Conversations | Month 3
  Patient participation in cost conversations is defined as percentage of patients in intervention arm participating in the scheduled conversation to discuss OOP.
Minutes of Patient Engagement in Cost Conversations | Month 3
  Patient engagement in cost conversations is defined as time (in minutes) that participants in the intervention arm spent discussing OOP cost with the financial counselor.
Patient Adherence to Cost Optimization Program | Month 3
  Patient adherence to cost optimization program is defined as the percentage of completed monthly contacts that participants in intervention arm have with study financial counselor.
Change in Utilization of Financial Supportive Services | Baseline, Month 3
  Use of financial supportive services will be assessed by asking participants if they received any assistance with paying for medication, imaging, or transportation to health provider visits in the past three months. For any financial support received, participants will be asked how they were linked to assistance. This is a qualitative assessment which does not provide a summary score.
Accuracy of OOP Cost Estimates | Month 3
  Accuracy of OOP cost estimates provided to patients in the intervention arm will be assessed by comparing the estimates to the amount stated in received medical bills, in a subset of patients who received medical bills.

OTHER OUTCOMES:
Change in Comprehensive Score for Financial Toxicity (COST) Questionnaire Score | Baseline, Month 3
  Financial toxicity is assessed using the COST questionnaire. The COST questionnaire includes 12 items asking how important specific financial scenarios are to participants on a scale of 0 to 4 where 0 = not at all and 4 = very much. Total scores will be calculated using responses from the first 11 items and range from 0 to 44. Certain items are reverse scored so that lower scores indicate greater financial toxicity.
Change in Cost-related Care Non-adherence | Baseline, Month 3
  Participants will be asked if they have forgone or delayed treatment or monitoring visits (e.g., medication, treatment other than prescribed medication, office visits, lab and imaging) related to MS in the last 3 months due to cost. Participants respond with "yes" or "no" and there is not a summary score for this assessment.
Change in Financial Hardship | Baseline, Month 3
  Participants will be asked about any financial hardship they are experiencing due to bills and income related to MS treatment. Participants will report if they had to change living situations, withdraw money from retirement or savings accounts, or if they had changes in income since their diagnosis, or had to obtain loans to pay medical bills. This is a qualitative assessment without a summary score.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Score | Baseline, Month 3
  Self-reported changes in physical, mental and social health will be assessed with the PROMIS Global Health instrument. This instrument includes 9 items scored from 1 to 5, where 1 is equivalent to poor health and 5 is equivalent to excellent health, plus a tenth item asking respondents to rate their average pain on a scale from 0 (no pain) to 10 (worst pain). Total score for the first 9 items range from 9 to 45 where higher scores indicate greater self-reported health. PROMIS t-scores will be calculated.
Change in Coping Behaviors | Baseline, Month 3
  Participants will be asked about any coping behaviors that were needed, such as decreased basic spending on food/clothing, decreased spending on leisure activities, or missed physician visits, due to bills related to MS treatment. This is a qualitative assessment without a summary score.
Change in Financial Self-Efficacy Scale (FSES) Score | Baseline, Month 3
  The FSES is a 6-item instrument assessing how confidently respondents can manage financial concerns. Responses to items are on a 4 point scale where 1 = exactly true and 4 = not at all true. Total scores range from 6 to 24 where higher scores indicate greater financial self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Sadigh, MD, Principal Investigator — Emory University
Locations (1):
- Neurology Clinic, 12 Executive Park Drive, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the manuscript (including text, tables, figures, and appendices) will be made available for sharing, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available for sharing beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be available to be shared with researchers who provide a methodologically sound proposal in order to achieve aims in the approved proposal. Proposals should be directed to gsadigh@emory.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Owens GM. Economic burden of multiple sclerosis and the role of managed sare organizations in multiple sclerosis management. Am J Manag Care. 2016 Jun;22(6 Suppl):s151-8. PMID 27356024
- [Background] Adelman G, Rane SG, Villa KF. The cost burden of multiple sclerosis in the United States: a systematic review of the literature. J Med Econ. 2013;16(5):639-47. doi: 10.3111/13696998.2013.778268. Epub 2013 Mar 7. PMID 23425293
- [Background] Himmelstein DU, Thorne D, Warren E, Woolhandler S. Medical bankruptcy in the United States, 2007: results of a national study. Am J Med. 2009 Aug;122(8):741-6. doi: 10.1016/j.amjmed.2009.04.012. Epub 2009 Jun 6. PMID 19501347
- [Background] Hartung DM, Bourdette DN, Ahmed SM, Whitham RH. The cost of multiple sclerosis drugs in the US and the pharmaceutical industry: Too big to fail? Neurology. 2015 May 26;84(21):2185-92. doi: 10.1212/WNL.0000000000001608. Epub 2015 Apr 24. PMID 25911108
- [Background] Rumrill PD Jr, Roessler RT, McMahon BT, Hennessey ML, Neath J. Gender as a differential indicator of the employment discrimination experiences of Americans with multiple sclerosis. Work. 2007;29(4):303-11. PMID 18057570
- [Background] de Souza JA, Yap B, Ratain MJ, Daugherty C. User beware: we need more science and less art when measuring financial toxicity in oncology. J Clin Oncol. 2015 Apr 20;33(12):1414-5. doi: 10.1200/JCO.2014.59.4986. Epub 2015 Mar 2. No abstract available. PMID 25732158
- [Background] Altice CK, Banegas MP, Tucker-Seeley RD, Yabroff KR. Financial Hardships Experienced by Cancer Survivors: A Systematic Review. J Natl Cancer Inst. 2016 Oct 20;109(2):djw205. doi: 10.1093/jnci/djw205. Print 2017 Feb. PMID 27754926
- [Background] de Souza JA, Yap BJ, Hlubocky FJ, Wroblewski K, Ratain MJ, Cella D, Daugherty CK. The development of a financial toxicity patient-reported outcome in cancer: The COST measure. Cancer. 2014 Oct 15;120(20):3245-53. doi: 10.1002/cncr.28814. Epub 2014 Jun 20. PMID 24954526
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] Streeter SB, Schwartzberg L, Husain N, Johnsrud M. Patient and plan characteristics affecting abandonment of oral oncolytic prescriptions. J Oncol Pract. 2011 May;7(3 Suppl):46s-51s. doi: 10.1200/JOP.2011.000316. PMID 21886519
- [Background] Lizan L, Comellas M, Paz S, Poveda JL, Meletiche DM, Polanco C. Treatment adherence and other patient-reported outcomes as cost determinants in multiple sclerosis: a review of the literature. Patient Prefer Adherence. 2014 Dec 4;8:1653-64. doi: 10.2147/PPA.S67253. eCollection 2014. PMID 25525341
- [Background] Benito-Leon J. Multiple sclerosis: is prevalence rising and if so why? Neuroepidemiology. 2011;37(3-4):236-7. doi: 10.1159/000334606. Epub 2011 Nov 30. No abstract available. PMID 22133765
- [Background] Jensen S, Given B. Fatigue affecting family caregivers of cancer patients. Support Care Cancer. 1993 Nov;1(6):321-5. doi: 10.1007/BF00364970. PMID 8156250
- [Background] Shankaran V, Leahy T, Steelquist J, Watabayashi K, Linden H, Ramsey S, Schwartz N, Kreizenbeck K, Nelson J, Balch A, Singleton E, Gallagher K, Overstreet K. Pilot Feasibility Study of an Oncology Financial Navigation Program. J Oncol Pract. 2018 Feb;14(2):e122-e129. doi: 10.1200/JOP.2017.024927. Epub 2017 Dec 22. PMID 29272200
- [Background] Rosenkrantz AB, Sadigh G, Carlos RC, Silva E 3rd, Duszak R Jr. Out-of-Pocket Costs for Advanced Imaging Across the US Private Insurance Marketplace. J Am Coll Radiol. 2018 Apr;15(4):607-614.e1. doi: 10.1016/j.jacr.2017.12.010. Epub 2018 Feb 22. PMID 29477290
- [Derived] Sadigh G, Coleman D, Lava N, Switchenko J, Vargas D, Duszak R Jr, Carlos RC. Patient-Specific Out-of-Pocket Cost Communication and Remote Financial Navigation in Patients with Multiple Sclerosis: A Randomized Controlled Feasibility Study. Mult Scler Relat Disord. 2022 Jun;62:103797. doi: 10.1016/j.msard.2022.103797. Epub 2022 Apr 10. PMID 35429820